CLINICAL TRIAL: NCT00501813
Title: A Randomized Controlled Trial of Multimodality Therapy in the Treatment of Palliative Resectable Hepatocellular Carcinoma With Intrahepatic Vessels Invasion
Brief Title: Multimodality Therapy for Palliative Resectable Hepatocellular Carcinoma With Intrahepatic Vessels Invasion
Acronym: MDTforHCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Cancer Center, Sun Yat-sen University, Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hcc-002
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Intrahepatic vessels invasion; Hepatectomy; Transcatheter arterial chemoembolization; Local regional treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery (Active Comparator): initial palliative hepatectomy followed by TACE and/or local regional treatment
  Interventions: Procedure: Hepatectomy
- no surgery (Experimental): TACE combined with local regional treatment without hepatectomy
  Interventions: Procedure: TACE combined with local regional therapies without hepatectomy

INTERVENTIONS:
Procedure: Hepatectomy — irregular Hepatectomy
  Arms: surgery
Procedure: TACE combined with local regional therapies without hepatectomy — TACE combined with RFA, MCT, PEI, and so on.
  Other Names: TACE combined with local regional treatment without hepatectomy
  Arms: no surgery

SUMMARY:
The purpose of this study is to compare the effects of different multimodality therapy strategies (initial hepatectomy followed by transcatheter hepatic arterial chemoembolization and/or local regional treatments compare with transcatheter hepatic arterial chemoembolization combined local regional treatments without hepatectomy)in the treatment of palliative resectable hepatocellular carcinoma with intrahepatic vessels invasion.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common neoplasm and the third cause of cancer-related death. At initial diagnosis, surgical resection is considered a potentially curative modality for HCC[1, 2], with the five-year survival rates for resectable patients 50-60%, however, only about 15% of patients have resectable disease and post-operative recurrence is common, remaining the main obstacle to long-term survival. On the one hand, the reason may be the multicentric genesis of HCC or the preoperatively micrometastasis that can not be resected during operation. Shi M, et al [3] reported that the appropriate resection margin was >= 2cm. The Liver Cancer Study Group of Japan (LCSGJ) defined[4]: absolute curative resection included liver resection with 1 cm of free surgical margin in patients with solitary tumor <= 2cm; relative curative resection included liver resection without 1 cm of free surgical margin but with the excised tumor tissue in patients with solitary tumor <= 2cm or liver resection with 1 cm of free surgical margin in patients with tumor >= 2cm (in either instance, no tumor thrombus may remain in the portal vein, hepatic vein, or bile duct in images of the remnant liver); relative non-curative resection, in which all macroscopic tumor tissue is removed; and absolute non-curative resection, which is liver resection with part of the macroscopic tumor tissue remaining. Either overall survival rates (OS) or disease-free survival rates (DFS) of HCC patients are higher in curative resection than in non-curative resection[4]. According to this definition, when the giant tumor located in middle liver, tumor with lymph nodes adjacent to abdominal aorta metastasis, multiple lesions (>= 3) or tumor with intrahepatic vessels invasion, the surgery will be non-curative. On the other hand, post-operative adjuvant therapy is one of the most effective treatment strategies in improving the survival rates of HCC patients[5]. Unfortunately, only about 15 randomized controlled trials have been reported on the post-operative adjuvant therapy until now. Most of them were single center, little sample clinical trials.

Recently, a series of studies have been reported that transcatheter arterial chemoembolization (TACE) is effective in HCC[6, 7]. Best results are seen in patients with small tumors and good liver function and 1 year survival has been shown to be of 30-50%. A recent meta-analysis showed a significant benefit of chemo-embolization with improvement in two-year survival[6]. TACE is one of most important therapy strategies on HCC. The 2007' NCCN clinical practice guidelines in oncology has included the TACE throughout the treatment guideline of unresectable HCC or resectable HCC (for some reason, hepatectomy was not carried out) or adjuvant therapy post-operative. But there are still lack of RCT studies.

In the patients with palliative resectable HCC, the presence of intrahepatic vessels invasion was usually regarded as the symbol of cancer cells hematogenous dissemination, which is associate with short-term recurrence and worse survival. For this special group patients, some authors insisted that aggressive therapy strategy-initial palliative hepatectomy followed by TACE and/or local regional treatments was most effective to prolong the survival of patients.While other authors,however,believed that too aggressive therapy was not best choice for these patients because of the suppression of immune system after palliative hepatectomy may potentially accelerate the growth of residual cancer cells. A relative conservative strategy-transcatheter hepatic arterial chemoembolization combined local regional treatments without hepatectomy should be used. The optimal therapy strategies are still in controversial.Only the multiple-center, great sample clinical RCT studies can answer this question[8]. The purpose of this study is to compare the effects of different multimodality therapy strategies (initial hepatectomy followed by transcatheter hepatic arterial chemoembolization and/or local regional treatments compare with transcatheter hepatic arterial chemoembolization combined local regional treatments without hepatectomy)in the treatment of palliative resectable hepatocellular carcinoma with intrahepatic vessels invasion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and <=70 years of age.
* Patients with palliative resectable HCC (all macroscopic tumor tissue can be removed), which have been histologically or cytologically documented. Documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable at screening.
* Patients must have at least one lesion that meets both of the following criteria:

  * The lesion can be accurately measured in at least one dimension according to RECIST (Section 10.7).
  * The lesion has not been previously treated with local therapy (such as surgery, radiation therapy, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation).
* Patients must have the tumor in the liver with intrahepatic vessels(portal vein/hepatic vein/bile duct) invasion, but all the tumor can be macroscopically removed.
* Patients who have an ECOG PS of 0 or 1.
* Cirrhotic status of Child-Pugh class A only. Child-Pugh status should be calculated based on clinical findings and laboratory results during the screening period.

Exclusion Criteria:

* Patient compliance is poor.
* The blood supply of tumor lesions is absolutely poor or arterial-venous shunt that TACE can not be performed.
* The vessels invasion beyond the following extent:

  * the main branch of portal vein;
  * the inferior vena cava;
  * the common hepatic duct.
* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted.
* History of cardiac disease:

  * congestive heart failure > New York Heart Association (NYHA) class 2;
  * active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted);
  * cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers, calcium channel blocker or digoxin;
  * uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of 3 antihypertensive drugs).
* Active clinically serious infections (> grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0).
* Known history of human immunodeficiency virus (HIV) infection.
* Known Central Nervous System tumors including metastatic brain disease.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Distantly extrahepatic metastasis.
* History of organ allograft.
* Drug abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial.
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
* Excluded therapies and medications, previous and concomitant:

  * Prior use of any systemic anti-cancer treatment for HCC, eg. chemotherapy, immunotherapy or hormonal therapy (except that hormonal therapy for supportive care is permitted). Antiviral treatment is allowed, however interferon therapy must be stopped at least 4 weeks prior randomization.
  * Prior use of systemic investigational agents for HCC
  * Autologous bone marrow transplant or stem cell rescue within four months of start of study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 1-, 3- and 5-year

SECONDARY OUTCOMES:
Quality of live | 1- and 3- month

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Qing Li, MD, Principal Investigator — Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University; Rong-Ping Guo, MD, Study Director — Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University
Locations (1):
- Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University,, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Arii S, Yamaoka Y, Futagawa S, Inoue K, Kobayashi K, Kojiro M, Makuuchi M, Nakamura Y, Okita K, Yamada R. Results of surgical and nonsurgical treatment for small-sized hepatocellular carcinomas: a retrospective and nationwide survey in Japan. The Liver Cancer Study Group of Japan. Hepatology. 2000 Dec;32(6):1224-9. doi: 10.1053/jhep.2000.20456. PMID 11093728
- [Background] Mise K, Tashiro S, Yogita S, Wada D, Harada M, Fukuda Y, Miyake H, Isikawa M, Izumi K, Sano N. Assessment of the biological malignancy of hepatocellular carcinoma: relationship to clinicopathological factors and prognosis. Clin Cancer Res. 1998 Jun;4(6):1475-82. PMID 9626465
- [Background] Shi M, Zhang CQ, Zhang YQ, Liang XM, Li JQ. Micrometastases of solitary hepatocellular carcinoma and appropriate resection margin. World J Surg. 2004 Apr;28(4):376-81. doi: 10.1007/s00268-003-7308-x. Epub 2004 Mar 17. PMID 15022021
- [Background] Ikai I, Arii S, Kojiro M, Ichida T, Makuuchi M, Matsuyama Y, Nakanuma Y, Okita K, Omata M, Takayasu K, Yamaoka Y. Reevaluation of prognostic factors for survival after liver resection in patients with hepatocellular carcinoma in a Japanese nationwide survey. Cancer. 2004 Aug 15;101(4):796-802. doi: 10.1002/cncr.20426. PMID 15305412
- [Background] Lau WY, Yu SC, Lai EC, Leung TW. Transarterial chemoembolization for hepatocellular carcinoma. J Am Coll Surg. 2006 Jan;202(1):155-68. doi: 10.1016/j.jamcollsurg.2005.06.263. Epub 2005 Oct 19. No abstract available. PMID 16377509
- [Background] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] Lopez PM, Villanueva A, Llovet JM. Systematic review: evidence-based management of hepatocellular carcinoma--an updated analysis of randomized controlled trials. Aliment Pharmacol Ther. 2006 Jun 1;23(11):1535-47. doi: 10.1111/j.1365-2036.2006.02932.x. PMID 16696801